CLINICAL TRIAL: NCT01132040
Title: An Open Label, Balanced. Randomized, Two-treatment, Two-period, Two-sequence, Single Dose,Crossover, Bioequivalence Study of Primidone 50 mg Tablets of Comparing With That of Mysoline® 50 mg Tablets Under Fasting Conditions.
Brief Title: Bioequivalence Study of Primidone Tablets 50 mg of Dr. Reddy's Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Mr. Indu Bhushan / Sr. Director - R&D, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P-620/06
Record Dates: First submitted 2010-05-26; First posted 2010-05-27 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2010-05

CONDITIONS: Healthy
Keywords: Bioequivalence; Crossover; Primidone
MeSH Terms: interventions — Primidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Primidone (Experimental): Primidone Tablets, USP 50 mg of Dr. Reddy's Laboratories
  Interventions: Drug: Primidone
- Mysoline (Active Comparator): Mysoline Tablets of Yamanouchi Pharma Technologies Inc,
  Interventions: Drug: Primidone

INTERVENTIONS:
Drug: Primidone — Primidone Tablets, USP 50 mg of Dr. Reddy's Laboratories Limited
  Other Names: Mysoline

SUMMARY:
The purpose of this study is to assess the bioavailability of Primidone 50 mg tablets of Dr.Reddy's comparing with that of Mysoline@ tablets of Yamanouchi Pharma Technologies Inc, in healthy, adult, human subjects under fasting conditions.

DETAILED DESCRIPTION:
An open label, balanced. randomized, two-treatment, two-period, two-sequence, single dose,crossover, bioequivalence study of Primidone 50 mg tablets of Dr.Reddy's Laboratories Limited, Generics, India comparing with that of Mysoline (containing Primidone 50 mg) tablets of Yamanouchi Pharma Technologies Inc, Norman, OK in healthy, adult, human subjects under fasting conditions with a washout period of 14 days.

ELIGIBILITY:
Inclusion Criteria:

Subjects must fulfill all of the following criteria to be considered for inclusion into this study:

1. Subjects who will provide written informed consent.
2. Subjects must be healthy, adult, human beings within 18-45 years of age (both inclusive)weighing at least 50 kg.
3. Having a Body Mass Index (BMI) between 18.5 and 24.9 (both inclusive), calculated as weight in Kg/height in m2
4. Subjects must be of normal health as determined by medical history and physical examination performed within 21 days prior to the commencement of the study.
5. Subjects whose screening laboratory values are within normal limits or considered by the physician/investigator to be of no clinical significance.
6. Availability of the subject for the entire study period and willingness to adhere to the protocol requirements as evidenced by written informed consent.

Exclusion Criteria:

The subjects will be excluded based on the following criteria during screening and during the study

1. Subjects incapable of understanding the informed consent.
2. Subjects who have:

   1. Systolic blood pressure less than 90 mm ofHg or more than 140 mm of Hg
   2. Diastolic blood pressure less than 60 mm of Hg or more than 94 mm of Hg. Minor deviations (2-4 mm of Hg) at check-in may be acceptable at the discretion of the physician/investigator.
   3. Pulse rate below 50/min or above 100/min.
3. History of hypersensitivity or idiosyncratic reaction to study drug or any other related drugs.
4. Any evidence of impairment of renal, hepatic, cardiac, lung or gastrointestinal function.
5. Consumption of grapefruit for the past ten days prior to the dosing day until the completion of the study.
6. Regular smoker who has a habit of smoking more than nine cigarettes per day and has difficulty in abstaining from smoking from 48 hours before dosing and during sampling period.
7. Subjects who have taken over the counter or prescribed medications and enzyme modifying or any systemic medication for during the last 7 and 30 days respectively before dosing.
8. Subjects who have participated in any other clinical investigation using experimental drug/donated blood in past 90 days before the date of start of study.
9. Subjects with clinically significant abnormalities (such as Laboratory Findings, ECG, X-Ray,Drugs of abuse, Alcohol etc.,) and/or with significant diseases (such as HIV, Hey, Syphilis,Hepatitis B etc.,).
10. Female subjects who are pregnant or who are able (women with child bearing potential) to become pregnant during the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2006-08; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax and AUC parameters | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Mohanlal shiva prasad sayana, Principal Investigator — Bioserve Clinical Research Pvt. Ltd., Hyderabad, A.P.
Locations (1):
- Bioserve Clinical Research Pvt. Ltd,, HYD, Andhra Pradesh, India